CLINICAL TRIAL: NCT04804215
Title: Intraductal Transanastomotic Stent in Duct-to-duct Biliary Reconstruction in Liver Transplantation: Multicenter, Randomized Controlled Trial
Brief Title: Intraductal Transanastomotic Stent in Duct-to-duct Biliary Reconstruction in Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Ho Joong Choi, Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Liver-01
Record Dates: First submitted 2021-03-07; First posted 2021-03-18 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Liver Transplant; Complications
Keywords: biliary reconstruction; Intraductal transanastomotic stent

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group in Intraductal transanastomotic stent (Experimental): Inclusion criteria
  * 19 years old or older ~ under 70 years old
    * Patients eligible for liver transplantation ③ Patients who have consented to written consent
  Intraductal transanastomotic stent was used during biliary reconstruction
  Interventions: Procedure: Intraductal transanastomotic stent group
- The controled group in non-Intraductal transanastomotic stent (Experimental): Inclusion criteria
  * 19 years old or older ~ under 70 years old
    * Patients eligible for liver transplantation ③ Patients who have consented to written consent
  No stent was used during biliary reconstruction
  Interventions: Procedure: No stent group

INTERVENTIONS:
Procedure: Intraductal transanastomotic stent group — When bile duct anastomosis is performed, a intraductal transanastomotic stent is inserted into the bile duct.
  Arms: The experimental group in Intraductal transanastomotic stent
Procedure: No stent group — Do not insert a stent into the bile duct during anastomosis of the bile duct.
  Arms: The controled group in non-Intraductal transanastomotic stent

SUMMARY:
Liver transplant surgery has been used as a major treatment modality for end-stage liver disease, hepatocellular carcinoma and acute liver failure due to innovations in surgical treatment of donors and recipients over the past decade. However, despite these advances, biliary tract complications are considered the technical "Achilles tendon" of liver transplantation because of their high incidence, long-term interventions and potential risk of transplant failure. The incidence of biliary tract complications after liver transplantation is still a high incidence, with a prevalence of 10-50% despite increasing technology and experience worldwide. Biliary tract complications are typically biliary tract leakage and biliary stricture, which are the cause of post-transplant morbidity and transplant loss. Most of the bile leakage occurs within 3 months after surgery, and the incidence of these early complications reaches 10-20%. Biliary stricture is a late complication that usually occurs within 5-8 months and can occur up to 1 year. The incidence of biliary stricture currently reported is still occurring in 5-30% of large clinical studies.

The use of external T-tubes to reduce biliary tract complications has been discussed for many years, and many published studies show no difference in biliary tract complications regardless of the use of T-tubes, as well as T-tube-related cholangitis and tube removal. Showed a relationship with certain morbidity rates, such as bile leakage.

Insertion of a stent into the bile duct has the advantage of preventing biliary complications while avoiding the side effects associated with the use of external T-tubes. We presented a preliminary study of 100 patients and confirmed that intrabiliary stents reduced biliary tract complications, and not using an intrabiliary stent was an independent risk factor for biliary stenosis.

Therefore, in this study, the purpose of this study was to determine the effective and rational use of intrabiliary stents through a randomized clinical trial according to the use of intrabiliary stents during biliary reconstruction in patients with liver transplant surgery. In addition, it is expected that clinical usefulness has not been announced until now in Korea, since a double-blind prospective randomized controlled clinical trial was conducted according to the presence or absence of an intrabiliary stent during biliary reconstruction in liver transplantation.

DETAILED DESCRIPTION:
Aim of study

1. Primary end-point To compare and evaluate the incidence of biliary tract complications within 6 months after surgery according to the presence or absence of an intrabiliary stent during biliary reconstruction in liver transplantation.
2. Second end-point Postoperative complications related to intrabiliary stent (cholangitis, acute pancreatitis, intestinal perforation, bleeding, etc.), liver transplantation and 6-month survival rate, hospitalization period, re-hospitalization, non-biliary complications, and liver through comparative analysis The purpose of this study is to check the clinical effectiveness of the use of an intrabiliary stent during transplantation.

Subject selection criteria, exclusion criteria, number of target subjects and their rationale

1. Selection criteria ① 19 years old or older ~ under 70 years old

   * Patients eligible for liver transplantation

     * Patients who have consented to written consent
2. Exclusion criteria

   * When performing hepato-plant anastomosis due to anatomical/biliary tract disease ② Patients who are not eligible for liver transplantation
3. Target number of people and basis for calculation Since this study was compared with the control group, the number of subjects was calculated using a non-inferiority test. To calculate the number of study subjects, in the existing literature, the incidence of surgical site infection was 1.33% in the group with antibiotics and 3.36% in the group without antibiotics. The difference between the ratio between the two groups is 2.02% larger in the test group than in the control group, and as a result of calculating the study subjects by assuming the upper limit of the confidence interval between the two groups as the non-inferiority margin of 5.4%, 72 subjects per each group were required, 10%. When calculating the dropout rate, 80 subjects per group, a total of 160 subjects, are required.

Study design

1. Clinical trial design This clinical trial is an exploratory clinical trial evaluating the safety and effectiveness of the use of intrabiliary stents during surgery in liver disease requiring transplantation. A screening test is performed on subjects who voluntarily agreed to participate in the trial in writing. On the day of surgery, after determining whether the selection/exclusion criteria are met, appropriate subjects are randomly assigned to the test group and the control group at a 1:1 ratio. In the control group, during bile duct anastomosis, a stent is not inserted into the bile duct, and the test group is inserted into the bile duct.

   On the OP day and on the discharge day, adverse reaction investigations, laboratory tests, and physical tests are conducted for safety and efficacy evaluation to evaluate postoperative pain and hospital stay. At one week after discharge from the hospital, adverse reactions, laboratory tests, and physical examinations are performed through an outpatient visit to evaluate the occurrence of postoperative complications related to infection, complications other than infection, and the need for additional procedures. In addition, the degree of postoperative pain, re-hospitalization, complications other than infection, and the need for additional procedures are evaluated and compared when visiting the emergency room due to the occurrence of postoperative infection-related complications within one month after discharge.
2. Target registration and randomization method Subjects who agreed to voluntarily participate in the trial after hearing the explanation about this clinical trial will be given a subject identification code in the order in which they signed the consent form at the screening visit.In this clinical trial, the comparability of the treatment group is maximized and the treatment group's Randomization is performed to ensure the scientific validity of the clinical trial by not involving the subjectivity of the investigator in the assignment.

   Block randomization is performed to divide the patients who satisfy the selection/exclusion criteria and agree to participate in the clinical trial into 2 groups and allocate them at a 1:1 ratio. For randomization, a statistical expert independent from this clinical trial generates a random assignment number using SAS ver.9.4 (SAS Institute Inc, NC, Cary, USA) or higher for Microsoft Windows and assigns it sequentially.
3. Operation and storage of random allocation In this clinical trial, randomization is operated by a third party, and the investigator receives subject consent from the subject during the screening period, and records necessary matters and test findings to determine the subject selection/exclusion criteria. At this time, the subjects will be given screening numbers in order.

   Finally, whether or not to participate in the clinical trial is determined by checking the suitability of the subject's clinical trial. Subjects who are determined to participate in the clinical trial are enrolled in the clinical trial and assigned a randomization number through a randomization envelope according to the randomization method to the test group or control group on the day of surgery, and based on the randomization table operated by the investigator (surgeon). Groups are allocated according to the subject assignment number.
4. Blind and unblind This clinical trial is a single-blind clinical trial. It should not be known to which group the subjects are assigned according to the assignment number, and the randomization table is kept by a third party, and the assigned envelope is managed in a separate place. During the clinical trial period, if blindfolding is required before the completion of the clinical trial due to a serious adverse reaction, the research manager contacts the randomization staff to review and approve the reason for the blindfolding, and then proceed with the blindfolding procedure.

Criteria for end of study and early termination

1. Criteria for cancellation and dropout In the case of the following occurrences, the clinical trial may be canceled or eliminated.

   ① When the subject requests to stop the test

   ② When the investigator judges that it is difficult to continue the clinical trial due to a serious adverse reaction

   ③ In case of violation of selection/exclusion criteria or serious violation of clinical trial plan

   ④ If the subject's follow-up observation is unsuccessful

   ⑤ When other testers decide that the test should be stopped
2. Treatment at the time of cancellation and dropout If a subject is discontinued or eliminated from the clinical trial, the investigator shall record the date of discontinuation and dropout, the reason for the discontinuation and dropout, and the treatment and progress at the time of discontinuation and dropout, along with all data acquired until the time of discontinuation and dropout. Subjects with early discontinuation in the clinical trial for any reason are not replaced.

Study method

1. Clinical trial intervention plan

   * Test group: stent insertion into the bile duct. (silastic stent)
   * Control: No stent insertion into the bile duct. Only subjects who have consented to participate in the clinical trial and have been randomly assigned to meet the criteria for selection/exclusion will perform the procedure.
2. Observation and inspection items

   * Written consent and demographic survey, physical measurements, vital signs Before entering the clinical trial, the investigator explains in detail the purpose and contents of this clinical trial to the subject and obtains written consent. After written consent, demographic information is investigated in the case record, and the date of written consent, subject's initials, gender, date of birth, etc. are recorded, and physical measurements (height, weight, BMI) and vital signs (systolic blood pressure, diastolic blood pressure, pulse, body temperature) Also measure and record. After each visit, physical measurements (weight, BMI) and vital signs (systolic blood pressure, diastolic blood pressure, pulse, and body temperature) are also measured and recorded.

     * Investigation of medical history and drug administration history At the screening visit, the interview and past medical records are reviewed, and the subject's entire life history is investigated and recorded based on the screening visit. In addition, after investigating and recording all drugs taken from 30 days prior to the screening visit, and checking whether there is a change in the condition of administration of the combination drug that was investigated during the screening test at each visit thereafter, and whether there is a new combination drug, Record it on the case record.

       * Physical and laboratory tests Physical and laboratory tests (blood and urine tests) are performed through screening visits and interviews at that visit, and the test results and normality are recorded in the case report.

         ④ ASA class According to the physical condition classification system established by the American Society of Anesthesiology, an evaluation is made between 1 and 6 points according to the physical condition of the patient undergoing surgery and anesthesia and recorded in the case report.

         ⑤ Imaging examination investigation Imaging tests should be collected if there are any results.

         ⑥ Surgery, hospitalization information investigation The following items are investigated for information on surgery and hospitalization.

         • Anesthesia time from start to finish

         • Operation time from abdominal incision to skin suture

         • Surgery time required for resection
         * Bleeding and intraoperative blood transfusions:

           -Measured in cc, taking into account the amount of blood inhaled during surgery and the weight of tape and gauze.
           * The amount of red blood cells and whole blood administered during surgery is measured in cc.
         * After surgery, the investigator evaluates the patient's recovery status (when the gas is released) once a day.
         * Evaluation items for patient recovery status: Record the progression of meals once a day every day, and if discharge is not made, the record of the progression of meals and postoperative complications on the discharge date is finally evaluated.

           * Investigation of complications related to infection Infection-related complications are divided into surgical site infection and wound infection, and other complications are investigated as non-infection-related complications. Symptoms such as fever are not collected as complications, but the cause is investigated and classified as complications. In addition, if additional procedures are needed due to the occurrence of related complications, the information should be collected.
3. Inspection items for each visit

   * Visit 1 (Screening, -28D ~ pre OP) • written consent

     * Determination of conformity to the selection/exclusion criteria
     * Demographic information and medical history survey
     * Physical examination
     * Physical measurement/Vital signs
     * Pre-drug investigation
     * ASA class
     * Abdominal ultrasound
     * Laboratory tests
     * Imaging examination investigation
     * Evaluation of pain level (VAS score)

       * Visit 2 (Baseline, OP day, surgery day)
     * Determination of conformity to the selection/exclusion criteria
     * Physical examination
     * Physical measurement/Vital signs
     * ASA class
     * Surgery Information Survey
     * Investigation of complications related to infection
     * Random assignment
     * Clinical trial intervention

       * Visit 3 (post OP±1D, discharge date)
     * Physical examination
     * Physical measurement/Vital signs
     * Concomitant drug investigation
     * ASA class
     * Laboratory tests
     * Hospitalization information investigation
     * Investigation of complications related to infection

       ④ Visit 4 (1W±1D)
     * Physical examination
     * Physical measurement/Vital signs
     * Concomitant drug investigation
     * ASA class
     * Hospitalization information investigation
     * Investigation of complications related to infection

       ⑤ Unscheduled visit (when visiting the emergency room) (OP+30D)
     * Hospitalization information investigation
     * Investigation of complications related to infection
     * Adverse reaction evaluation

ELIGIBILITY:
Inclusion Criteria:

* 19 years old or older ~ under 70 years old

  * Patients eligible for liver transplantation ③ Patients who have consented to written consent

Exclusion Criteria:

① When performing hepato-plant anastomosis due to anatomical/biliary tract disease

② Patients who are not eligible for liver transplantation

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of biliary tract complications within 6 months after surgery | 6 months
  The incidence of biliary tract complications within 6 months after surgery according to the presence or absence of an intrabiliary stent during biliary reconstruction in liver transplantation

SECONDARY OUTCOMES:
Postoperative complications rate (%) related to intrabiliary stents | 6 months
  Postoperative complications rate (%) related to intrabiliary stents (cholangitis, acute pancreatitis, intestinal perforation, bleeding, etc.), liver transplantation
6-month survival rate | 6 months
  6-month survival rate (%)
hospitalization period | 21days
  length of hospital stay (days)
re-hospitalization rate | 6 months
  re-hospitalization rate (%)
non-biliary complications rate | 6 months
  non-biliary complications rate (%) such as atelectasis, pneumonia, wound infection, sepsis, septic shock, etc.
Clinical effectiveness of biliary stent use | 6 months
  the need for additional procedures rate (%) such as endoscopic intervention or angiography

CONTACTS AND LOCATIONS:
Overall Officials: Yoonkyung Woo, MD, Study Director — Seoul St. Mary's Hospital; Yoonyung Choi, MD, Study Director — Seoul St. Mary's Hospital; Jin Ha Chun, MD, Study Director — Seoul St. Mary's Hospital
Locations (1):
- Department of HBP Surgery, Seoul St. Mary's hospital, Seoul, Seocho-gu, Banopo-dong, South Korea

IPD SHARING:
Plan to Share IPD: No